CLINICAL TRIAL: NCT02791035
Title: Correlation Between Change of HbA1c, Urinary Glucose Excretion and Other Factors in Patients Treated With Ipragliflozin
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Collaborators: Severance Hospital (Other); Samsung Medical Center (Other); Kyung Hee University Hospital at Gangdong (Other); Astellas Pharma Korea, Inc. (Industry)
Responsible Party: Principal Investigator, WOO JE LEE, Associate Professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AMC 2016-0100
Record Dates: First submitted 2016-05-27; First posted 2016-06-06 (Estimated); Last update posted 2017-07-05 (Actual); Status verified 2017-07

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

ARMS (1):
- Ipragliflozin (Experimental): Ipragliflozin 50 mg/tablet, orally, 1 tablet once daily for 12 weeks
  Interventions: Drug: Oral administration of Ipragliflozin

INTERVENTIONS:
Drug: Oral administration of Ipragliflozin

SUMMARY:
The purpose of this study is to examine the correlation between change of HbA1c, urinary glucose excretion and other factors when ipragliflozin is added to preexisting therapy in subjects with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Subject who has written informed consent
* Subjects who are diagnosed as type 2 diabetes mellitus
* Subjects who are 20 to 70 years old
* Subjects on a stable diet and exercise at least 8 weeks prior to the study participation
* Stable doses of the following medications for 8 weeks or more but, HbA1c level of 7.0 to 9.5% (Metformin, Metformin + SU, Metformin + DPP-4 inhibitor, Metformin + TZD, TZD, TZD + SU, TZD + DPP-4 inhibitor, SU, SU + DPP-4 inhibitor, DPP-4 inhibitor)

Exclusion Criteria:

* Type 1 DM
* Gestational DM
* Diabetic ketoacidosis
* CKD stage 3B-5 (eGFR 45)
* Severe infection, serious trauma, or perioperative period
* Known or suspected hypersensitivity to ipragliflozin
* Symptomatic urogenital infection
* Chemotherapy or radiation therapy for malignant tumor or diagnosis of malignant tumor within 5 years (except for thyroid cancer)
* Under the therapeutic intervention and/or another clinical study using IP drug
* Hepatic disease ( 3 times of upper normal limit of AST or ALT)
* Serious voiding difficulty due to neurogenic bladder or prostate hyperplasia
* Drugs not allowed for concomitant use

  * Alpha glucosidase inhibitor or meglitinide within 60 days prior to screening
  * Insulin within 60 days prior to screening
  * Systemic steroid use (PO, IV or IM) over 2 weeks within 3 months prior to screening
  * Inhalation or pleural intracavitary injection of steroid known as having high systemic absorption rate
* GLP-1 agonist (except for exenatide) within 60 days prior to screening
* Heart failure (NYHA class III-IV) or uncontrolled arrhythmia within 6 months prior to screening
* Cardiovascular diseases (unstable angina, myocardial infarction, transient ischemic attack, cerebrovascular disease, coronary artery bypass graft, or percutaneous coronary intervention) within 3 months prior to screening
* Subjects who are not eligible to the study according to an investigator's decision
* Inability to read the consent form
* Pregnancy, lactation, or plan to get pregnant during the study period

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-06; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Correlation between change of HbA1c and urinary glucose excretion | Baseline and week 12

SECONDARY OUTCOMES:
Correlation between reduction in HbA1c and various parameters (HOMA-IR, HOMA-ß, insulinogenic index) | Baseline and week 12
Correlation between increase in urinary glucose excretion and various parameters (HOMA-IR, HOMA-ß, insulinogenic index) | Baseline and week 12
Change of HbA1c | Baseline and week 12
Chang e of fasting glucose | Baseline and week 12
Change of waist circumference | Baseline and week 12
Percentage of subjects achieving the target HbA1c(<6.5%) | week 12

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea